CLINICAL TRIAL: NCT03004391
Title: Development of a Decision Aid to Facilitate Ovarian Cancer Patient's Choices Regarding Biomarker CA125
Status: Completed | Type: Observational
Sponsor: Vejle Hospital (Other)
Collaborators: Danish Cancer Society (Other); Design School Kolding (Other)
Responsible Party: Sponsor
Other Study IDs: CA125-DA
Record Dates: First submitted 2016-12-15; First posted 2016-12-28 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Ovarian Cancer
Keywords: Shared decision making; Follow-up
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In 2015 the Danish Health authorities initiated major changes in the national follow-up (FU) program for ovarian cancer patients. The new FU program argues that there is no effect of routine monitoring of tumour marker CA125. Now every patient needs to choose if they wish routine measurement of CA 125 to be part of the follow-up program.

Shared Decision Making (SDM) can help health professionals develop a more individualized care plan in collaboration with the patient, as stated in the revised national FU program. Due to the complexity and challenges within ovarian cancer care, this is an evident area of focus.

SDM is defined as an approach in which the clinician and patient go through all phases of the decision-making process together and share the preference for treatment and reach an agreement on treatment choice. Clinicians have information about disease, tests and treatments, whereas patients hold information about their life circumstances, goals of life, and preferences for healthcare. SDM thereby offers a way of individualizing recommendations, according to patients' special needs and preferences. SDM has potential to give the patients a higher quality of healthcare by putting the patient in the center of care.

Decision aids (DA) are tools that can provide information and systematically describe the advantages and disadvantages of a specific intervention or monitoring, which can help patients become involved in decision making. Using evidence-based DA leads to improvement in knowledge, better understanding of screening, prevention and treatment options, and more accurate perception of risks for the patients.

All participants fill in a demographic and Decisional Conflict Scale questionnaire at baseline. After having been presented with the decision aid and made a choice as to CA125, the participants will complete the CollaboRATE and Decisional Conflict Scale questionnaire dealing with confidence as to the choice made and the level of shared decision making experienced. Six months later the Decision Regret Scale questionnaire is to be completed to reveal any regrets in relation to the CA125 decision.

For a preliminary investigation of the applicability of the DA, 15-20 patients not eligible for this study will be asked for their opinion.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Histologically confirmed epithelial ovarian, fallopian tube or serous primary peritoneal cancer
* Have completed their first line treatment, with complete remission.
* Manage to read and speak Danish

Exclusion Criteria:

* Have recurrent disease after first line treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Patient uncertainty as to routine measurement of CA125 is measured by combined questionnaires CollaboRATE and Decisional Conflict Scale. | 6 months

SECONDARY OUTCOMES:
Patient satisfaction as to choice made measured by questionnaire Decision Regret Scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anette S. Kargo, MD, Principal Investigator — University of Southern Denmark and Vejle Hospital, Denmark; Karina D. Steffensen, MD, PhD, Study Director — University of Southern Denmark and Vejle Hospital, Denmark
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark